CLINICAL TRIAL: NCT02066038
Title: A Multi-center, Open-labeled Phase 2 Study of First Line Intermittent and Maintenance of Erlotinib in Combination With Pemetrexed/Carboplatin in ⅢB/IV Non Small Cell Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Mutation
Brief Title: Intermittent and Maintenance of Erlotinib in Combination With Pemetrexed/Carboplatin in Ⅲb/IV Non Small Cell Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, LongHao, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-FXY-025
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Lung, Carcinoma
Keywords: chemotherapy; maintenance therapy; erlotinib
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Pemetrexed 500mg/m2+Carboplatin area under curve(AUC)=5, every 3 weeks, maximum 4 cycles, Erlotinib 150mg/d every cycle d2-15, and Erlotinib 150mg/d from the last cycle until disease progression
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 150mg po on days 2-15 of each 3 week cycle for 4 cycles and 150mg po per day after 4 cycles until disease progression
  Other Names: Tarceva

SUMMARY:
EGFR-tyrosine kinase inhibitor(TKI)- ie, erlotinib, gefitinib, has been recommended as the first option for EGFR-mutated IIIb/IV NSCLC by serial trials as it prolonged patients' progression-free survival. The OPTIMAl trial indicated that those who received TKI and chemotherapy during the whole treatment window survived longest. Unfortunately, previous studies(INTACT, TRIBUTE et al) that concurrently combined TKI and cytotoxic regimens failed to improve survival in unselected patients. To avoid the potential synergistic antagonism, the FAST-ACT II trial committed a sequential strategy and find a superiority in the combination arm upon chemotherapy even in EGFR-mutated group. However, pharmaceutically, the continuous administration of an EGFR-TKI before subsequent chemotherapy in FAST-ACT II could obviate the effects of cytotoxic agents due to the erlotinib-induced G1 arrest.

On the basis of these and other studies, the investigators hypothesized that a better sequential combination strategy of EGFR-TKI and chemotherapy (adding a EGFR-TKI wash-out window before chemotherapy) would be more efficacious than chemotherapy alone. In this study, the investigators investigate the efficacy(PFS:progression free survival), safety, and adverse-event profile of chemotherapy plus intermittent and maintenance of erlotinib, when these drugs were used as first-line treatment in who had non-squamous lung carcinoma with EGFR gene mutation in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age.
* Present with histologically proven or cytological diagnosis of non-Squamous NSCLC Stage IIIB or IV as defined by the American Joint Committee on Cancer Staging Criteria for Lung Cancer, that is not amenable to curative therapy,such as surgery or radiotherapy and so on.
* No prior systemic chemotherapy or targeted therapy for lung cancer before screening.
* Confirmed activating mutation of EGFR-ie, an exon 19 deletion or an exon 21 L858R point mutation.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1.
* Adequate organ function.
* Prior radiation therapy allowed to <25% of the bone marrow . Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study enrollment. Patients must have recovered from the acute toxic effects of the treatment prior to study enrollment.
* Signed informed consent document on file.
* Estimated life expectancy of ≥12 weeks.
* Patient compliance and geographic proximity that allow adequate follow up.

Exclusion Criteria:

* Known severe hypersensitivity to erlotinib.
* Patients with uncontrolled brain metastasis.
* Pleural effusion or pericardiac effusion that cannot be controlled by drainage or other procedures.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Interstitial pneumonia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-04 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors(RECIST) 1.1 | eight weeks
  Patients were imaged with computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Overall Officials: Hao Long, Prof, Principal Investigator — Sun Yat-sen University